CLINICAL TRIAL: NCT02615925
Title: Descriptive Study of Mental Activity in the Emergency Department of the Centre Hospitalier de Mayotte
Brief Title: Descriptive Study of Mental Activity
Acronym: URGPSYMAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9417; 2014-A00807-40 (Other: RCB number)
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Psychiatric Disorder Requiring Hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psychiatry Consultation (Other): Psychiatry Consultation, it is proposed by one of the investigators, patients that clinical data from this psychiatric examination, conducted as part of their usual care, are recorded as part of the research that their is proposed and explained. An information note is then distributed and not collected their opposition
  Interventions: Other: Psychiatry Consultation

INTERVENTIONS:
Other: Psychiatry Consultation — Psychiatry Consultation

SUMMARY:
Provide a description of patients admitted in the psychaitric department of the Mayotte Hospital

DETAILED DESCRIPTION:
This feature and the proximity of Mayotte with developing countries give this department different specificities, both culturally and medically. Indeed, the local population of lifestyle and specific beliefs, combining Islam and animism. Thus, a person with mental suffering is traditionally treated by a wizard who will come into contact with the spirits that inhabit the person, the community that supports the patient remains at home.

Mayotte is far behind compared to the metropolis where the supply of psychiatric care with a fragile population, a care network being created, and few downstream solutions To handle crisis situations, emergency unit and psychiatric liaison, speaking to general emergencies was established in 2010. It is currently the only access to emergency psychiatric care on the island.

The situations covered by this unit are for patients of all ages and all social and geographical origins, reflecting the demographics of the population.

Investigator has only quantitative data (number of patients / year) and has no qualitative analysis tool. No epidemiological research has been done to date in this direction.

The aim of our study was to analyze the impact of various psychiatric disorders represented Mayotte of the emergency hospital to get a statistical picture of its business.

This description will present to the scientific community the specifics of this department

ELIGIBILITY:
Inclusion Criteria:

Patient in need of psychiatric care in the emergency department

Exclusion Criteria:

* Patient leaves the emergency department against medical advice or fugue
* Patient leaves the service without the medical diagnosis is made
* Patient in exclusion period determined by a previous search
* Patients for whom it is impossible give clear information
* Patient who manifested their opposition to participate in research
* Patient minor whose parental agreement has been reached
* Patient on safeguarding justice whose guardian will not be contacted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

PRIMARY OUTCOMES:
Describe the mental activity | 1 day
  Describe the mental activity of the emergency hospital of Mayotte (clinical observations obtained during routine psychiatric consultation) That is to say, describe the different psychiatric pathologies of all patients presenting to the emergency department of CH Mayotte.

SECONDARY OUTCOMES:
Estimated incidence rates of various psychiatric pathologies | 1 day
  Estimated incidence rates of various psychiatric pathologies (clinical observations obtained during routine psychiatric consultation)
Search factors associated with different pathologies | 1 day
  Search factors associated with different pathologies (clinical observations obtained during routine psychiatric consultation)
Creating a database for further research. | 1 day
  Creating a database for further research (clinical observations obtained during routine psychiatric consultation)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOLINARI, Principal Investigator — University Hospital of Montpellier, Montpellier, France, 34295
Locations (1):
- CH de MAYOTTE, Montpellier, Mamoudzou, France